CLINICAL TRIAL: NCT02163512
Title: Effect of Beta-adrenergic Blockers on Cardiac Function, Systemic and Splanchnic Haemodynamic and Kidney Function in Cirrhotic Patiets With Refractory Ascites
Acronym: ALB-BET
Status: Completed | Type: Observational
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Sponsor
Other Study IDs: ALB-BET-2011-01
Record Dates: First submitted 2014-06-10; First posted 2014-06-13 (Estimated); Last update posted 2019-02-11 (Actual); Status verified 2016-06

CONDITIONS: Hepatic Cirrhosis
Keywords: Hepatic cirrhosis; Ascites; Beta blockers treatment
MeSH Terms: conditions — Liver Cirrhosis; Ascites

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Non-refractory ascites
- Refractory ascites

SUMMARY:
Multicentric, observational and prospective study with two groups of treatment: Refractory ascites and non-refractory ascites. All patients should be prescribed beta-adrenergic blockers as primary or secondary profilaxis for variceal bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80
* Patients previously prescribed with beta-blockers
* Any type of hepatic cirrosis that has been diagnosed by clinical, analytic and image criteria
* Mild to serious ascites. Classification on refractory or non-refractory ascites depends on the patient´s response to diuretic treatment. Refractory ascites is defined by the Ascites´Board International Criteria as the lack of response, ascites recurrency or complications occurrence by diuretic drugs uptake
* Esophageal varicose vein in which beta blockers treatment is indicated as primary or secondary prophylaxis. Primary prophylaxis is indicated for big esophageal varicose veins, small varicose veins with red signs or varicose veins in patients with B-C Child-Pugh stage. Secondary prophylaxis is indicated for all those patients that have previously presented varicose bleeding.
* Patients giving a written consent to participate in the study after having received enough information about the design, objectives and risks.

Exclusion Criteria:

* Hepatocellular carcinoma >5 cm
* Total portal vein thrombosis or Cavernous transformation of the portal vein
* Insuficiencia renal (creatinina sérica >3 mg/dl).
* Kidney insufficiency (seric creatinine >3 mg/dl)
* Contraindications to beta-blockers: Cardiac or breathing insufficiency, auricular-ventricular blocking grade >1.
* Anticoagulant treatment
* Patients with a intrahepatic portosystemic shunt
* Beta-blockers Hypersensitivity
* Pregnancy and breastfeeding
* Women of childbearing age must commit to undergo an effective contraception during the treatment and at least one month after finishing it.
* Patients with severe controlled or not controlled psychiatric condition
* Patients´ lack of commitment to follow all visits.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hepatic cirrhoris and refractory or non-refractory ascites. These patients are going to be treated with beta blockers as primary or secondary prophylaxis of variceal bleeding
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2014-03-12 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Cardiac function | Baseline and after 4 weeks
  * Echocardiography: changes in left ventricular ejection fraction, cardiac output,
  * Electrocardiography: changes in Qt interval
Kidney function | Baseline and after 4 weeks
  * Echocardiography: Renal vascular Doppler ultrasonographic parameters (resistive index of kidney arteries)
  * Blood test: serum creatinine, estimated glomerular filtration rate (eGFR) calculated by the Modification of Diet in Renal Disease formula, IL18, KIM1, NGAL

SECONDARY OUTCOMES:
Inflammatory markers and vasoactive endogenous system | Baseline and after 4 weeks
  * Levels of monoaminergic systems: variations in activity of the autonomous nervous system (levels of renin, aldosterone and noradrenaline)
  * Immune system activation: TNF-alpha, IL 6, TNFR I y II, LBP

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid

REFERENCES:
- [Derived] Tellez L, Ibanez-Samaniego L, Perez Del Villar C, Yotti R, Martinez J, Carrion L, Rodriguez de Santiago E, Rivera M, Gonzalez-Mansilla A, Pastor O, Bermejo J, Banares R, Albillos A. Non-selective beta-blockers impair global circulatory homeostasis and renal function in cirrhotic patients with refractory ascites. J Hepatol. 2020 Dec;73(6):1404-1414. doi: 10.1016/j.jhep.2020.05.011. Epub 2020 May 21. PMID 32446716